CLINICAL TRIAL: NCT01056601
Title: Phase II Study of Panobinostat (LBH589) Given in Combination With Bortezomib (Velcade) in Patients With Pancreatic Cancer Progressing on Gemcitabine Therapy Alone or Gemcitabine in Combination
Brief Title: Panobinostat & Bortezomib in Pancreatic Cancer Progressing on Gemcitabine Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding not available
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009LSUC012; X05302 (Other: Millennium Pharmaceuticals, Inc.)
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Results first posted 2011-08-26 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-11

CONDITIONS: Pancreatic Cancer
Keywords: insulinoma; cancer of pancreas; neoplasms, pancreas; alpha-cell tumor; glucagonoma; beta-cell tumor; somatostatinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Insulinoma; Glucagonoma; Somatostatinoma | interventions — Bortezomib; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pancreatic Cancer Patients (Experimental): Pancreatic cancer patients who received treatment with bortezomib and panobinostat after progressing on gemcitabine.
  Interventions: Drug: Bortezomib; Drug: Panobinostat

INTERVENTIONS:
Drug: Bortezomib — 1.3 mg/m^2 administered intravenously twice daily on days 1 and 8 for 2 weeks followed by 10 day rest period
  Other Names: Velcade
Drug: Panobinostat — 20 milligrams administered orally 3 times weekly for 2 weeks on Days 1,3,5,8,10 and 12 followed by 9 day rest period
  Other Names: LBH589

SUMMARY:
Cancer results from multiple mutations which cause cells to grow uncontrolled. It therefore may be necessary to inhibit several oncogenic targets to affect cancer cell growth. Studies have shown that panobinostat (LH589) causes a wide range of effect on endothelial cells that lead to inhibition of tumor angiogenesis (a fundamental step in the transition of tumors from a dormant state to a malignant one). Bortezomib triggers cell death in pancreatic cancer cells but the mechanism is not well defined but has been determined to be cytostatic. Combining these two drugs may work together in the treatment of pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of locally advanced or metastatic pancreatic cancer (except neuroendocrine tumors, but including ampullary cancer) with progression after standard first line therapy that included gemcitabine (single agent or combination)
* Measurable disease on computated tomography (CT) scan per Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* At least 28 days from previous systemic therapy, including investigational agents and 1st dose of study treatment and recovered from any acute toxic effects of that treatment before study enrollment.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 - Ability to provide written consent
* Must meet hematology and biochemistry laboratory criteria within 14 days of study enrollment:

  * Neutrophil count >1500/mm^3
  * Platelet count >100,000/mm^L
  * Hemoglobin > or = 9 g/dL
  * Aspartate aminotransferase (AST/SGOT) or Alanine transaminase (ALT/SGPT) < or = 2.5 times upper limit of normal (ULN)or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement
  * Serum bilirubin < or = 1.5 x ULN
  * Serum creatinine < or = 1.5 x ULN or 24-hour creatinine clearance ≥ 50 ml/min
  * Total serum calcium (corrected for serum albumin) or ionized calcium ≥ lower limit of normal (LLN)
  * Serum phosphorus > or = LLN
  * Serum potassium > or = LLN
  * Serum sodium ≥ LLN
  * Serum magnesium ≥ LLN
  * Serum albumin ≥ LLN or 3g/dl
  * Patients with any elevated Alkaline Phosphatase due to bone metastasis can be enrolled
* Baseline multi gated acquisition scan (MUGA) or echocardiogram (ECHO) must demonstration left ventricular ejection fraction (LVEF) > or = 50%
* Normal thyroid function within normal limits. Note: Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
* Women of childbearing potential (WOCBP) must have a negative pregnancy tests within 7 days of study treatment administration and willing to use 2 methods of contraception

Exclusion Criteria:

* > 1 prior systemic treatment regimen for pancreatic cancer
* Prior histone deacetylase (HDAC), deacetylase (DAC), heat shock protein 90 (HSP90) inhibitors or valproic acid for treatment of cancer
* Anyone needing valproic acid for any medical condition during the study or 5 days prior to panobinostat treatment
* Impaired cardiac function

  * Complete left bundle branch block or use of a permanent cardiac pacemaker, congenital long QT syndrome, history or presence of ventricular tachyarrhythmias, clinically significant resting bradycardia (<50 beats per minute), QTcF > 450 msec on screening ECG, or right bundle branch block + left anterior hemiblock (bifascicular block)
  * Presence of atrial fibrillation (ventricular heart rate >100 bpm)
  * Previous history angina pectoris or acute myocardial infarction (MI) within 6 months of study enrollment
  * Congestive heart failure (New York Heart Association functional classification III-IV) or baseline MUGA/Echo shows LVEF < 50%
* Uncontrolled hypertension defined as hypertensive blood pressure of SBP > 140 or DBP > 90, despite antihypertensive medications
* History of deep vein thrombosis (DVT), pulmonary emboli or other blood clotting abnormality within 3 months of study enrollment
* Ongoing need for anti-coagulation therapy except daily low dose aspirin (≤ 100 mg/day) or low molecular weight heparin
* Concomitant use of drugs with risk of causing torsades de pointes
* Anyone with unresolved diarrhea > or = grade 2 at time of enrollment
* Impairment of gastrointestinal function or disease that may significantly alter the absorption of panobinostat
* Grade 2 or greater peripheral neuropathy within 14 days of enrollment
* Serious concomitant medical or psychiatric disorders (e.g., active infection, uncontrolled diabetes)
* Patients who have received chemotherapy, any investigational agent or undergone major surgery < 4 weeks prior to starting study drug
* Male patients whose sexual partners are WOCBP and not using double method of contraception during the study and 3 months following.
* Known positivity for human immunodeficiency virus (HIV) or hepatitis C
* Hypersensitivity to bortezomib, boron or mannitol History of another primary malignancy within 5 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arkadiusz Dudek, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pancreatic Cancer Patients: Pancreatic cancer patients who received treatment with bortezomib (1.3 mg/m^2 administered intravenously twice daily on days 1 and 8 for 2 weeks followed by 10 day rest period) and panobinostat (20 milligrams administered orally 3 times weekly for 2 weeks on Days 1,3,5,8,10 and 12 followed by 9 day rest period) after progressing on gemcitabine.
Period: Overall Study
Arm/Group | Pancreatic Cancer Patients
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pancreatic Cancer Patients
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Median number of months before disease progressed in patient on gemcitabine when treated with the combination of panobinostat and bortezomib. Progression free survival is measured from randomization until the subject has documented disease progression by an objective measure. Subjects must be alive with no more than 20% increase in tumor size to qualify for progression free survival. Changes in tumor size are defined by RECIST criteria.
Time Frame: Up to 1 Year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pancreatic Cancer Patients
Number analyzed (Participants) | 7
Months | 2.1 [1.7 to 2.3]

2. Secondary Outcome: Number of Participants by Tumor Response
Description: Number of patients whose tumor has responded to study therapy is determined using Response Evaluation Criteria In Solid Tumors. Progressive Disease (PD) is assessed if the sum of the diameters has increased by ≥ 20% and ≥ 5 mm from nadir (including baseline if it is the smallest sum). Objective response is measured by tumor reduction as defined in the RECIST criteria. Tumor shrinkage must be at least 30% to qualify as an objective response.
Time Frame: Up to 1 Year
Measure: Number; unit: Participants
Arm/Group | Pancreatic Cancer Patients
Number analyzed (Participants) | 7
Participants
  Progressive Disease | 5
  No data available | 2
  Objective Response | 0

3. Secondary Outcome: Duration of Response
Description: Duration of response is calculated as (Date of First Disease Progression or Death as a Result of any Cause whichever Comes First - Date of First Objective Status Assessment of Confirmed Complete or Partial Response as defined by RECIST criteria).
Time Frame: Up to 1 Year
Measure: Number; unit: Weeks
Arm/Group | Pancreatic Cancer Patients
Number analyzed (Participants) | 7
Weeks | 0

ADVERSE EVENTS:
Time Frame: Overall Study
Arm/Group | Pancreatic Cancer Patients
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pancreatic Cancer Patients (N=7)
Dehyration (Metabolism and nutrition disorders) | 1 (1)
Fever (General disorders) | 1 (1)
INR Increased (Investigations) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pancreatic Cancer Patients (N=7)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 5 (6)
Anorexia (Gastrointestinal disorders) | 2 (2)
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorder, other (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Creatinine increased (Renal and urinary disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (Endocrine disorders) | 2 (2)
Eye disorder, other (Eye disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
GGT increased (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Renal and urinary disorders) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 7 (10)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (Gastrointestinal disorders) | 3 (3)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Study was terminated early leading to small numbers of subjects analyzed; no solid conclusion can be derived.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes